CLINICAL TRIAL: NCT00100126
Title: A Phase III, Investigator Blind, Randomized, Multicenter Study to Evaluate the Efficacy and Safety of APC-231 Sprinkle QD for 7 Days vs Penicillin VK 10 mg/kg QID for 10 Days in Pediatric Patients With Streptococcus Pyogenes
Brief Title: APC-231 Once a Day (QD) for 7 Days vs. Penicillin Taken Four Times a Day (QID) in Pediatric Patients With Strep Throat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advancis Pharmaceutical Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 231.301
Record Dates: First submitted 2004-12-23; First posted 2004-12-24 (Estimated); Last update posted 2006-10-25 (Estimated); Status verified 2005-04

CONDITIONS: Pharyngitis
Keywords: Pharyngitis; Strep throat
MeSH Terms: conditions — Pharyngitis

INTERVENTIONS:
Drug: Amoxicillin Pulsatile Release Multiparticluate Sprinkle

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of APC-231 QD for 7 days in the bacteriological outcome at the Test of Cure Visit.

ELIGIBILITY:
Inclusion Criteria:

Give informed consent, assent, and documentation of patient authorization for disclosure of study results.

Since all patients are below the legal age of consent, assent from the patient must be obtained (as applicable following state regulations) and written informed consent obtained from the parent or legal guardian.

* Age > = 6 months -12 years.
* A clinical diagnosis of acute tonsillitis and/or pharyngitis defined as having the clinical signs and symptoms compatible with tonsillitis and/or pharyngitis, including sore throat or difficulty feeding or swallowing or irritability that suggests the presence of a sore throat with at least one of the following:

  * Tonsillar or pharyngeal exudate
  * Tender cervical lymph nodes
  * Fever or history of fever treated with antipyretics
  * Odynophagia
  * Uvular edema
  * Pharyngeal Erythema of moderate or greater intensity
  * Elevated white blood cell (WBC) >12,000/mm3 or 10% bands
  * Red tongue and prominent papillae (Strawberry tongue)
* A positive rapid screening test for S. pyogenes (enzyme immunoassay; SiGNIFY™ Strep A Test).
* Patient is an appropriate candidate for oral antibiotic therapy and can swallow the study dosage forms.
* Females must be non-lactating and:

  * If of childbearing potential and sexually active, the patient must have a negative prestudy urine pregnancy test and be utilizing acceptable birth control methods throughout the study.

Exclusion Criteria:

* Chronic or recurrent (two weeks duration two times per year) odynophagia or enlarged tonsils secondary to viral or proven bacterial etiology.

  * The need for hospitalization or I.V. antimicrobial therapy.
  * Pharyngitis known or suspected to be due to a pathogen resistant to beta-lactam antimicrobials.
  * Patients who are known carriers of S. pyogenes.
  * Previous allergy, serious adverse reaction to, or intolerance to, penicillin or any other member of the beta-lactam class of antimicrobials.
  * Any serious illness or concomitant condition that the investigator judges would preclude the study evaluations or make it unlikely that the course of study therapy and follow-up could be completed. This would also include:
* Any rapidly progressive underlying disease with a shortened life expectancy.
* The inability to swallow the study dosage form.
* Unable to understand the requirements of the study.
* Neutropenia (<1000 PMNs/mm3) or other known immunocompromised state.
* Hard chills or rigors.

  * Seizure disorder or lowered seizure threshold. This does not exclude children with previous febrile seizures.
  * Psychiatric condition requiring use of major tranquilizers.
  * Pregnancy or nursing.
  * Expectation that additional effective systemic antibacterials would be required for any condition during the duration of the study.
  * Current drug or alcohol abuse.
  * Receipt of any experimental drug or medical device within the previous 30 days (or are scheduled to receive any other experimental procedures during the study period).
  * Previous treatment under this protocol.
  * Systemic antimicrobial therapy with benzathine penicillin within 30 days or azithromycin within 14 days.
  * Hospitalization within the month prior to study admission, during which antibacterial therapy was administered.
  * The presence of clinically significant hematologic conditions or cardiac valvular disease.
  * History of cardiovascular disease, renal disease, or neurological disease secondary to previous infection with S. pyogenes.
  * Probenecid treatment or systemic steroids during the duration of the study.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500
Dates: Start 2004-12; Study Completion 2005-06

PRIMARY OUTCOMES:
Bacteriological outcome at Test of Cure Visit

SECONDARY OUTCOMES:
Bacteriological outcome at Late Post Therapy Visit
Clinical Outcomes
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Susan Clausen, PhD, Study Director — Advancis Pharmaceutical Corp
Locations (2):
- United States (2):
  - Simpsonville, South Carolina
  - Institute for Neuroscience Research, Salt Lake City, Utah